CLINICAL TRIAL: NCT04149470
Title: Proton Pump Inhibitor (PPI) Response in Eosinophilic Esophagitis Assessed by Transnasal Endoscopy (TNE)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1119
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE; PPI; Proton Pump Inhibitor; Omeprazole; eosinophil; TNE; Transnasal Endoscopy; Esophageal Diseases; Esophagitis; Gastrointestinal Diseases; Eosinophilia; Gastroenteritis; Eosinophilic Oesophagitis; Transnasal Esophagogastroduodenoscopy; Transnasal Esophagoscopy
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophageal Diseases; Esophagitis; Gastrointestinal Diseases; Eosinophilia; Gastroenteritis | interventions — Omeprazole; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Omeprazole (Experimental): Participants will receive high dose PPI therapy (Omeprazole 20mg twice daily) and will be evaluated for histological improvement.
  Interventions: Drug: Omeprazole 20mg BID

INTERVENTIONS:
Drug: Omeprazole 20mg BID — High dose PPI therapy (Omeprazole 20mg twice daily)

SUMMARY:
This study will enroll participants who have been diagnosed with Eosinophilic Esophagitis (EoE). Upon study enrollment, the participant will begin a proton pump inhibitor (PPI), Omeprazole 20mg twice daily. After taking Omeprazole for four weeks, the participant will have a Transnasal Endoscopy, and biopsies will be taken to determine the histological change. If the biopsies are abnormal, the participant continues Omeprazole and will undergo another endoscopy at eight weeks. The study aims to determine the percentage of children with Eosinophilic Esophagitis who improve with PPI use and to determine the length of time and effectiveness of PPI therapy in the management of EoE. The investigators hypothesize that following the initiation of PPI for treatment of Eosinophilic Esophagitis, biopsies obtained will show decreasing eosinophil counts at four weeks, which is sooner than the previously reported eight-week period.

DETAILED DESCRIPTION:
This study aims to learn more about the subset of children with Eosinophilic Esophagitis (EoE) who are on treatment with a proton pump inhibitor (PPI). EoE is an increasingly common allergic condition of the esophagus for which we have limited treatment options. This study will be helpful in evaluating the minimal time frame required for histological improvement with the use of high dose PPI. The study will enroll participants who have been diagnosed with Eosinophilic Esophagitis (EoE) and are recommended by their physician to begin PPI treatment with Omeprazole 20 mg twice daily. After taking Omeprazole for four weeks, the participant will undergo an unsedated Transnasal Endoscopy (TNE) in the outpatient clinic at Children's Hospital Colorado. TNE is a test in which the doctor inserts a skinny bendable tube with a camera through the nose to look directly into the esophagus (the tube connecting the mouth to the stomach when you swallow) and is an alternative method to assess esophageal mucosa without requiring general anesthesia. Biopsies will be collected during the TNE to determine if there is histological change. If the biopsies are normal, the participant will complete the study. If biopsies are abnormal, and EoE is still active, the participant will continue the Omeprazole and undergo the standard of care endoscopy at eight weeks. The participant will choose the type of endoscopy- unsedated TNE or esophagogastroduodenoscopy (EGD) under anesthesia. Participants will also complete surveys during study enrollment about medication compliance, Eosinophilic Esophagitis symptoms, anxiety, TNE experience, and undergo a physical exam. The investigators hypothesize that following the initiation of PPI for treatment of Eosinophilic Esophagitis, biopsies obtained will show decreasing eosinophil counts at four weeks, which is sooner than the previously reported eight-week period. Results from this study will be generalizable to the pediatric EoE population and the knowledge gained will provide key preliminary data to support clinical recommendations for pediatric EoE patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Male or female, ages 8-22
* Current diagnosis of Eosinophilic Esophagitis (≥ 15 eos/HPF) within the last 6 months
* Able to swallow pills or open capsule to take medication with apple sauce
* Weight >20kg
* Willing to undergo unsedated transnasal endoscopy (TNE)

Exclusion Criteria:

* Inability or unwillingness of participant to give written informed consent or comply with study protocol.
* Have a known bleeding disorder
* Current topical esophageal corticosteroid or systemic steroid treatment within past 8 weeks
* No therapy with H2 therapy within the past 16 weeks
* Planned or anticipated change in the diet during the study duration.
* Planned or anticipated change in other corticosteroid medications
* Uncontrolled cough, rhinorrhea, rhinitis obstructing nasal passages, GI illness or determination of significant illness at screening
* Pregnancy, breast feeding or plans to become pregnant
* Use of investigational drug within last 16 weeks
* Allergy to any medications used for procedures
* Allergy to PPI
* Past or current medical problems or findings from physical exam or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Histological Response at baseline | baseline
  The histological response will be based on pathologist's review of esophageal biopsies for pediatric participants with Eosinophilic Esophagitis (EoE). EoE diagnosis is identified if there are ≥ 15 eosinophils per high power field (hpf) in the esophagus.
Change in Histological Response Rate at four weeks | 4 weeks
  The histological response will be based on pathologist's review of esophageal biopsies for pediatric participants with Eosinophilic Esophagitis (EoE) who are prescribed a high dose proton pump inhibitor, Omeprazole 20 mg twice daily. Biopsies will be evaluated using the EoE histological scoring system. Response will be defined as the peak eosinophil count of < 15 eosinophils per high power field and normal will be defined at 0 eosinophils per high power field.
Change in Histological Response Rate at eight weeks | 8 weeks
  The histological response will be based on pathologist's review of esophageal biopsies for pediatric participants with Eosinophilic Esophagitis (EoE) who are prescribed a high dose proton pump inhibitor, Omeprazole 20 mg twice daily. Biopsies will be evaluated using the EoE histological scoring system. Response will be defined as the peak eosinophil count of < 15 eosinophils per high power field and normal will be defined at 0 eosinophils per high power field.

SECONDARY OUTCOMES:
PEESS (Pediatric Eosinophilic Esophagitis Symptom Severity Module) scores at enrollment | At enrollment
  The PEESS (Pediatric Eosinophilic Esophagitis (EoE) Symptom Scores) validated assessment tool will be completed by participant and parent at the enrollment visit. PEESS is a metric that seeks to capture EoE specific symptoms directly from children and their parents. Scores range from 0 (never) to 4 (almost always) and each question measures frequency and severity of EoE symptoms in the past month.
PEESS (Pediatric Eosinophilic Esophagitis Symptom Severity Module) scores at four weeks | 4 weeks
  The PEESS (Pediatric Eosinophilic Esophagitis (EoE) Symptom Scores) validated assessment tool will be completed by participant and parent after four weeks using Omeprazole 20mg twice daily. PEESS is a metric that seeks to capture EoE specific symptoms directly from children and their parents. Scores range from 0 (never) to 4 (almost always) and each question measures frequency and severity of EoE symptoms in the past month.
PEESS (Pediatric Eosinophilic Esophagitis Symptom Severity Module) scores at eight weeks | 8 weeks
  The PEESS (Pediatric Eosinophilic Esophagitis (EoE) Symptom Scores) validated assessment tool will be completed by participant and parent after eight weeks using Omeprazole 20mg twice daily. PEESS is a metric that seeks to capture EoE specific symptoms directly from children and their parents. Scores range from 0 (never) to 4 (almost always) and each question measures frequency and severity of EoE symptoms in the past month.
Eosinophilic Esophagitis Histology Scoring System (HSS) scores at enrollment | At enrollment
  The EoE HSS provides a method to objectively assess histology change in esophageal biopsies beyond eosinophil count. The HSS evaluates eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces (DIS), surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. The study pathologist will review the historical esophageal biopsies using the HSS.
Eosinophilic Esophagitis Histology Scoring System (HSS) scores at four weeks | 4 weeks
  The EoE HSS provides a method to objectively assess histology change in esophageal biopsies beyond eosinophil count. The HSS evaluates eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces (DIS), surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. The study pathologist will review the participant's esophageal biopsies collected after four weeks of Omeprazole 20mg twice daily using the HSS.
Eosinophilic Esophagitis Histology Scoring System (HSS) scores at eight weeks | 8 weeks
  The EoE HSS provides a method to objectively assess histology change in esophageal biopsies beyond eosinophil count. The HSS evaluates eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces (DIS), surface epithelial alteration, dyskeratotic epithelial cells, and lamina propria fibrosis. The study pathologist will review the participant's esophageal biopsies collected after eight weeks of Omeprazole 20mg twice daily using the HSS.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Nguyen, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Result] Friedlander JA, DeBoer EM, Soden JS, Furuta GT, Menard-Katcher CD, Atkins D, Fleischer DM, Kramer RE, Deterding RR, Capocelli KE, Prager JD. Unsedated transnasal esophagoscopy for monitoring therapy in pediatric eosinophilic esophagitis. Gastrointest Endosc. 2016 Feb;83(2):299-306.e1. doi: 10.1016/j.gie.2015.05.044. Epub 2015 Jul 2. PMID 26142551
- [Result] Nguyen N, Lavery WJ, Capocelli KE, Smith C, DeBoer EM, Deterding R, Prager JD, Leinwand K, Kobak GE, Kramer RE, Menard-Katcher C, Furuta GT, Atkins D, Fleischer D, Greenhawt M, Friedlander JA. Transnasal Endoscopy in Unsedated Children With Eosinophilic Esophagitis Using Virtual Reality Video Goggles. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2455-2462. doi: 10.1016/j.cgh.2019.01.023. Epub 2019 Jan 29. PMID 30708107
- [Result] Dellon ES, Gonsalves N, Hirano I, Furuta GT, Liacouras CA, Katzka DA; American College of Gastroenterology. ACG clinical guideline: Evidenced based approach to the diagnosis and management of esophageal eosinophilia and eosinophilic esophagitis (EoE). Am J Gastroenterol. 2013 May;108(5):679-92; quiz 693. doi: 10.1038/ajg.2013.71. Epub 2013 Apr 9. PMID 23567357
- [Result] Molina-Infante J, Ferrando-Lamana L, Ripoll C, Hernandez-Alonso M, Mateos JM, Fernandez-Bermejo M, Duenas C, Fernandez-Gonzalez N, Quintana EM, Gonzalez-Nunez MA. Esophageal eosinophilic infiltration responds to proton pump inhibition in most adults. Clin Gastroenterol Hepatol. 2011 Feb;9(2):110-7. doi: 10.1016/j.cgh.2010.09.019. Epub 2010 Oct 1. PMID 20920599
- [Result] Molina-Infante J, Bredenoord AJ, Cheng E, Dellon ES, Furuta GT, Gupta SK, Hirano I, Katzka DA, Moawad FJ, Rothenberg ME, Schoepfer A, Spechler SJ, Wen T, Straumann A, Lucendo AJ; PPI-REE Task Force of the European Society of Eosinophilic Oesophagitis (EUREOS). Proton pump inhibitor-responsive oesophageal eosinophilia: an entity challenging current diagnostic criteria for eosinophilic oesophagitis. Gut. 2016 Mar;65(3):524-31. doi: 10.1136/gutjnl-2015-310991. Epub 2015 Dec 18. PMID 26685124
- [Result] Dellon ES, Liacouras CA, Molina-Infante J, Furuta GT, Spergel JM, Zevit N, Spechler SJ, Attwood SE, Straumann A, Aceves SS, Alexander JA, Atkins D, Arva NC, Blanchard C, Bonis PA, Book WM, Capocelli KE, Chehade M, Cheng E, Collins MH, Davis CM, Dias JA, Di Lorenzo C, Dohil R, Dupont C, Falk GW, Ferreira CT, Fox A, Gonsalves NP, Gupta SK, Katzka DA, Kinoshita Y, Menard-Katcher C, Kodroff E, Metz DC, Miehlke S, Muir AB, Mukkada VA, Murch S, Nurko S, Ohtsuka Y, Orel R, Papadopoulou A, Peterson KA, Philpott H, Putnam PE, Richter JE, Rosen R, Rothenberg ME, Schoepfer A, Scott MM, Shah N, Sheikh J, Souza RF, Strobel MJ, Talley NJ, Vaezi MF, Vandenplas Y, Vieira MC, Walker MM, Wechsler JB, Wershil BK, Wen T, Yang GY, Hirano I, Bredenoord AJ. Updated International Consensus Diagnostic Criteria for Eosinophilic Esophagitis: Proceedings of the AGREE Conference. Gastroenterology. 2018 Oct;155(4):1022-1033.e10. doi: 10.1053/j.gastro.2018.07.009. Epub 2018 Sep 6. PMID 30009819
- [Result] Gutierrez-Junquera C, Fernandez-Fernandez S, Cilleruelo ML, Rayo A, Echeverria L, Quevedo S, Bracamonte T, Roman E. High Prevalence of Response to Proton-pump Inhibitor Treatment in Children With Esophageal Eosinophilia. J Pediatr Gastroenterol Nutr. 2016 May;62(5):704-10. doi: 10.1097/MPG.0000000000001019. PMID 26513622
- [Result] Lucendo AJ, Arias A, Molina-Infante J. Efficacy of Proton Pump Inhibitor Drugs for Inducing Clinical and Histologic Remission in Patients With Symptomatic Esophageal Eosinophilia: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2016 Jan;14(1):13-22.e1. doi: 10.1016/j.cgh.2015.07.041. Epub 2015 Aug 3. PMID 26247167
- [Result] Philpott H, Nandurkar S, Royce SG, Gibson PR. Ultrathin unsedated transnasal gastroscopy in monitoring eosinophilic esophagitis. J Gastroenterol Hepatol. 2016 Mar;31(3):590-4. doi: 10.1111/jgh.13173. PMID 26426817
- [Result] Dumortier J, Ponchon T, Scoazec JY, Moulinier B, Zarka F, Paliard P, Lambert R. Prospective evaluation of transnasal esophagogastroduodenoscopy: feasibility and study on performance and tolerance. Gastrointest Endosc. 1999 Mar;49(3 Pt 1):285-91. doi: 10.1016/s0016-5107(99)70002-7. PMID 10049409
- [Result] Yagi J, Adachi K, Arima N, Tanaka S, Ose T, Azumi T, Sasaki H, Sato M, Kinoshita Y. A prospective randomized comparative study on the safety and tolerability of transnasal esophagogastroduodenoscopy. Endoscopy. 2005 Dec;37(12):1226-31. doi: 10.1055/s-2005-921037. PMID 16329022